CLINICAL TRIAL: NCT04529629
Title: Precise Diagnosis, Treatment and Prognostic Evaluation of Complicated Adrenal Tumor Diseases
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Weiqing, PhD, MD, Shanghai Jiao Tong University School of Medicine
Other Study IDs: CCEMD-2020-0825
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Complicated Adrenal Tumor Diseases
MeSH Terms: interventions — Surgical Procedures, Operative; Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, Serum, plasma and full blood samples are retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- primary aldosteronism
  Interventions: Other: surgery or drug
- pheochromocytoma
  Interventions: Other: surgery or drug
- adrenocortical carcinoma
  Interventions: Other: surgery or drug

INTERVENTIONS:
Other: surgery or drug — pheochromocytoma and adrenocortical carcinoma need surgery and primary aldosteronism need drug according to the genetic results

SUMMARY:
The adrenal gland is an important organ that produces life hormones. There are many types of adrenal tumors, which tend to occur in young adults and affect the whole body. It has the dual threat: hormone secretion and tumor metastasis. At present, there are four major dilemmas in the clinical diagnosis and treatment of adrenal tumors: 1) Pulse secretion of the hormones, which are affected by many factors; and the diagnostic value of single hormone is limited; 2) Traditional imaging cannot accurately reflect the characteristics of hormone secretion. The prognosis cannot be accurately predicted; 3) The molecular characteristics of tumor cells and the microenvironment are unclear, making it difficult to implement early diagnosis and precise treatment; 4) Traditional pathology cannot determine the nature and long-term prognosis of the tumor, which makes the treatment delay, and the disease prognosis is extremely poor. It threatens the lives of patients.

Starting from solving the above-mentioned key problems in the early stage, the research team has systematically established new clinical diagnostic technologies, hormone dynamic tests to accurately assess hormone secretion and segmented blood collection hormone determination technologies to accurately locate adrenal tumors; A series of important research results have been published in Science, Lancet Diabetes & Endocrinology, Cell Research, etc To sum up, the goal of this research is improving the early diagnosis rate of complicated adrenal tumors especially in malignant tumors, developing the optimal treatment plan, avoiding unnecessary surgical treatment, improving the quality of life of patients, reducing mortality. This project will further integrate the adrenal cortex and medulla hormone mass spectrometry detection and the molecular markers of adrenal tumors through phenotypic, functional imaging, and molecular pathological evaluations, and built a sensitive drug screening platform that integrates visual drug response and molecular characteristics, thereby achieving precise diagnosis and treatment of complicated adrenal tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and ≤ 75 years
* Diagnosis of Patients with primary aldosteronism, pheochromocytoma, and cortical cancer
* Gender: males and females
* Provide written informed consent
* Satisfactory compliance

Exclusion Criteria:

1. Patients with renal insufficiency (Cr>2 times the upper limit of normal).
2. Patients with a history of liver cirrhosis.
3. Patients who are currently using corticosteroids.
4. Patients with cardiac insufficiency (NYHA cardiac function classification grade 3 and above or EF<50%).
5. Patients with stroke and acute myocardial infarction in the past 6 months.
6. Patients during pregnancy and lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Age ≥ 18 years old and ≤ 75 years
  * Diagnosis of Patients with primary aldosteronism, pheochromocytoma, and cortical cancer
  * Gender: males and females
  * Provide written informed consent
  * Satisfactory compliance
  Exclusion Criteria:
  1. Patients with renal insufficiency (Cr>2 times the upper limit of normal).
  2. Patients with a history of liver cirrhosis.
  3. Patients who are currently using corticosteroids.
  4. Patients with cardiac insufficiency (NYHA cardiac function classification grade 3 and above or EF<50%).
  5. Patients with stroke and acute myocardial infarction in the past 6 months.
  6. Patients during pregnancy and lactation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2040-08-30 (Estimated); Study Completion 2041-08-30 (Estimated)

PRIMARY OUTCOMES:
tumor biochemical marker treatment response | 20 years
  * Complete remission (normalization of tumor markers);
    * Partial remission (reduction of tumor markers ≥ 50%); ③No change (decrease of tumor markers <50% or increase ≤25%); ④Disease progression (tumor markers increased> 25%).
Tumor volume assessment: According to RECIST (version 1.1). | 20 years
  * Complete response: All target lesions disappear, and the short axis of any pathological lymph nodes must be reduced to <10 mm.
    * Partial Response: The total diameter of the target lesions is reduced by at least 30% compared with the baseline.
      * Progressive Disease: Take the minimum value of the sum of the diameters of all target lesions measured during the study as the reference, and the relative increase in diameter sum by at least 20% ④Stable Disease: Based on the minimum value of the sum of the diameters of all target lesions measured during the study, the reduction of the target lesion did not reach PR, and the degree of increase did not reach PD, between PR and PD.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided